CLINICAL TRIAL: NCT06174701
Title: Building Resilience for Surgical Recovery: Feasibility and Acceptability Pilot Study
Brief Title: Building Resilience for Surgical Recovery
Acronym: BRSR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Victoria Tang, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HSC-MS-24-0384; 5K76AG059931-05 (NIH)
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Psychosocial Functioning; Surgery; Older Adults; Physical Function; Postoperative Outcome; Depressive Symptoms
Keywords: Psychosocial Functioning; Surgery; Older Adults; Physical Function; Postoperative Outcome; Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The data collectors on the study team will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Problem Solving Therapy (PST) (Experimental): Participants in the intervention arm will receive Problem Solving Therapy (PST). Meetings via videoconferencing or phone will occur at a frequency of 1 time every week for an estimated 2-3 sessions before surgery and 6-7 sessions after surgery for a total of 9 sessions. Essential components of the PST that the patient will be taught include: (1) define the nature of the problem, (2) generate wide range of possible solutions, (3) systematically evaluate the potential solutions and select the most optimal ones to implement, and (4) monitor and evaluate the actual solution outcome after implementation.
  Interventions: Behavioral: Problem Solving Therapy (PST)
- Enhanced Usual Care (Experimental): Participants in the control arm will receive "enhanced usual care". They will receive additional mental health education in the form of educational handouts mailed or emailed to them.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Problem Solving Therapy (PST) — PST intervention in the form of one-on-one coaching in preparation for surgery and post-operative care. This coaching consists of educating and guiding the patient in developing problem-solving skills. Please refer to the PST Handbook for further detail on the therapy sessions.
  Arms: Problem Solving Therapy (PST)
Behavioral: Enhanced Usual Care — Participants in the control arm will receive "enhanced usual care". They will receive additional mental health education in the form of educational handouts mailed or emailed to them.
  Arms: Enhanced Usual Care

SUMMARY:
The goal of this clinical trial is to test problem solving therapy (PST) in older adults who are undergoing major surgery. The main question it aims to answer is: What is the feasibility and acceptability of delivering PST to older surgical patients with depressive symptoms or report lacking social support in the pre-operative and post-operative setting?

DETAILED DESCRIPTION:
A pilot test of a 9-session psychosocial intervention (Problem Solving Treatment, PST) will be conducted at the University of Texas, Southwestern Medical Center (UTSW). Ninety older surgical patients will be recruited from UTSW's Peri-operative Senior Health (POSH) clinic, with 20 for training, 35 randomized to the intervention arm, and 35 in the control arm. Preliminary data from this study will inform an R01 submission assessing the impact of PST on post-operative functional recovery.

Summary of Objectives:

1. Examine the feasibility of implementing an evidence-based psychosocial intervention, PST, for older surgical patients with depressive symptoms.
2. Demonstrate the acceptability of the intervention delivery for older surgical patients with depressive symptoms.
3. Evaluate the potential improvement in function and reduction in depressive symptoms.

Setting:

Ninety older adults undergoing major surgery will be recruited at the UTSW POSH clinic during the pre-operative period over a 6-month time frame. UTSW POSH sees 15-20 older surgical patients pre-operatively a week.

Recruitment and Enrollment:

Participants will be recruited through two pathways - clinician referral and self-referral. (1) Clinician referral: clinicians will refer via recruitment flyer, by the clinic team at the clinic visit, or via email to the study team. (2) Self-referral: recruitment flyers will be utilized in waiting rooms and clinical offices for interested patients to contact the study team.

Clinician Referral Details:

Clinicians will provide the research team with the patient's name and phone number for recruitment if they believe the patient is experiencing depressive symptoms and has a life expectancy of more than 6 months. The study team will reach out to the patient to recruit them into the study.

Enrollment and Consent:

Enrollment and consent will be conducted over the phone, and consent forms with DocuSign will be sent via email. To reduce discrimination against older adults unfamiliar with the technology, those unable to sign the consent form via DocuSign will be mailed the paper consent form with return postage to sign and send back. Consent will be stored in RedCAP.

Training of Interventionists:

Interventionists will undergo training with a problem-solving therapy master trainer. Participants will be recruited for this training until all interventionists meet criteria for intervention delivery. Refer to the training participant consent form for details.

ELIGIBILITY:
Inclusion criteria:

* ≥ 65 years of age on the day of surgery
* Scheduled major surgery with an anticipated hospital stay of 3+ days. Major operations include: orthopedic, thoracic or abdominal, cardiac procedures
* Depressive symptoms - Patient Health Questionnaire (PHQ-9) screening with a score of 5+, 5-9 being subclinical depression and scores up to 27 indicating increasing depression. If the score is 5-9, we need to have at least one of these items included: "at least one of the endorsed items needs to be depressed mood or diminished activities" (questions #1 and #2)

Exclusion criteria:

* Those with severe cognitive impairment - Short Portable Mental Status Questionnaire (SPMSQ) screening with a score of 5+ errors, 5-8 being moderate to severe cognitive impairment
* Unable to read, speak, and understand English
* Current alcohol or other substance abuse (scoring 2+ on CAGE questionnaire or answering yes to "Do you currently use any non-prescription drugs or substances?")
* Life expectancy is 6 months or less

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-06-04 (Estimated); Study Completion 2025-06-04 (Estimated)

PRIMARY OUTCOMES:
Functional Recovery as Assessed by Score on the World Health Organization Disability Assessment Schedule (Brief-WHODAS) | 6 months after baseline
  6-month functional recovery is measured by a comparison of the pre- and post-operative function using self-report to the World Health Organization Disability Assessment Schedule (Brief-WHODAS). Brief-WHODAS is a 12-item questionnaire where scores assigned to each of the items ["none" (0), "mild" (1), "moderate" (2), "severe" (3), and "extreme" (4)] are summed. The "summary score" is then converted into a metric ranging from 0 to 100 (where 0 = no disability; 100 = full disability). The rationale for using 6 months for follow-up is that after a major surgery, older adults can take up to 6 months to recover to their new functional baseline and has been used in previous studies.

SECONDARY OUTCOMES:
Depressive Symptoms as Assessed by Score on the by the Patient Health Questionnaire (PHQ-9) | 3 months and 6 months after baseline
  The secondary outcome is 3 and 6-month depressive symptoms, as measured by the Patient Health Questionnaire (PHQ-9). It is a 9-item questionnaire in which each item can be scored as 0 - Not at all, 1 - Several days, 2 - More than half the days, or 3 - Nearly every day. The total score is obtained by summing the scores for each of the nine items, resulting in a total score range from 0 to 27. 0 indicates no/minimal depression, and 27 indicates severe depression.

OTHER OUTCOMES:
Physical pain | Day of enrollment (baseline), 1 month after baseline, 3 months after baseline and 6 months after baseline.
  Brief Pain Inventory (BPI) (1 question from the 11 questions) - "Throughout our lives, most of us have had pain from time to time (such as minor headaches, sprains, and toothaches). Have you had pain other than these everyday kinds of pain today?" Yes to indicate pain and no to indicate no pain.
Cognition | Day of enrollment (baseline), 1 month after baseline, 3 months after baseline and 6 months after baseline.
  The Short Portable Mental Status Questionnaire (SPMSQ) (10-items) for assessment of cognitive function in older adults. Scoring scale of 0-8: Screening with a score of 5+ errors, 5-8 being moderate to severe cognitive impairment.
Depressive symptoms | Day of enrollment (baseline), 1 month after baseline, 3 months after baseline and 6 months after baseline.
  Measured by the Patient Health Questionnaire (PHQ-9), a 9-item self-report questionnaire assesses depression to gauge the severity of depression over the past two weeks. Screening with a score of 5+, 5-9 indicating subclinical depression and scores up to 27 indicating increasing depression. If the score is 5-9, at least one of these items needs to be included: "at least one of the endorsed items needs to be depressed mood or diminished activities" (questions #1 and #2).
Self-efficacy | Day of enrollment (baseline), 1 month after baseline, 3 months after baseline and 6 months after baseline.
  As measured by General Perceived Self-efficacy Scale (GSE). A 10-item questionnaire with the total score being the sum of the all items. Scores range from 0-40 with a higher score indicating more self-efficacy.
Anxiety | Day of enrollment (baseline), 1 month after baseline, 3 months after baseline and 6 months after baseline.
  As measured by General Anxiety Disorder (GAD-7). A 7-item questionnaire with a score of 0-4 indicating minimal anxiety; 5-9 indicating mild anxiety; 10-14 indicating moderate anxiety; 15-21 indicating severe anxiety. Anxiety will also be measured by the Behavioral Activation for Depression Scale Short Form (BADS-SF). A 9-item questionnaire with 6 items focusing on activation and 3 items focusing on avoidance. The range of scores is 0 to 54, with high scores representing higher activation.
Social Support | Day of enrollment (baseline), 1 month after baseline, 3 months after baseline and 6 months after baseline.
  As measured by Patient-Reported Outcomes Measurement Information System (PROMIS)- Emotional support and instrumental support questions. Scores for each set up questions range from 8-40 where 8 indicates no social support and 40 indicates social support. The initial collection will be used as the baseline measure against which subsequent collections will be compared.
Physical Function | Day of enrollment (baseline), 1 month after baseline, 3 months after baseline and 6 months after baseline.
  As measured by World Health Organization Disability Assessment Schedule 2.0 (Brief-WHODAS), as this is a community dwelling older adult population and this scales from activity of daily living (ADL) to participation in society. Brief-WHODAS is a 12-item questionnaire where scores assigned to each of the items - "none" (0), "mild" (1) "moderate" (2), "severe" (3) and "extreme" (4) - are summed. The "summary score" is them converted into a metric ranging from 0 to 100 (where 0 = no disability; 100 = full disability). Will also be measured by Katz Index of Independence in Activities of Daily Living (ADL) and Lawton Instrumental Activities of Daily Living Scale (IADL).

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Tang, MD, MAS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makary MA, Segev DL, Pronovost PJ, Syin D, Bandeen-Roche K, Patel P, Takenaga R, Devgan L, Holzmueller CG, Tian J, Fried LP. Frailty as a predictor of surgical outcomes in older patients. J Am Coll Surg. 2010 Jun;210(6):901-8. doi: 10.1016/j.jamcollsurg.2010.01.028. Epub 2010 Apr 28. PMID 20510798
- [Background] Oxman TE, Freeman DH Jr, Manheimer ED. Lack of social participation or religious strength and comfort as risk factors for death after cardiac surgery in the elderly. Psychosom Med. 1995 Jan-Feb;57(1):5-15. doi: 10.1097/00006842-199501000-00002. PMID 7732159
- [Background] Etzioni DA, Liu JH, O'Connell JB, Maggard MA, Ko CY. Elderly patients in surgical workloads: a population-based analysis. Am Surg. 2003 Nov;69(11):961-5. PMID 14627256
- [Background] Boyd CM, Landefeld CS, Counsell SR, Palmer RM, Fortinsky RH, Kresevic D, Burant C, Covinsky KE. Recovery of activities of daily living in older adults after hospitalization for acute medical illness. J Am Geriatr Soc. 2008 Dec;56(12):2171-9. doi: 10.1111/j.1532-5415.2008.02023.x. PMID 19093915
- [Background] Berian JR, Zhou L, Hornor MA, Russell MM, Cohen ME, Finlayson E, Ko CY, Robinson TN, Rosenthal RA. Optimizing Surgical Quality Datasets to Care for Older Adults: Lessons from the American College of Surgeons NSQIP Geriatric Surgery Pilot. J Am Coll Surg. 2017 Dec;225(6):702-712.e1. doi: 10.1016/j.jamcollsurg.2017.08.012. Epub 2017 Oct 17. PMID 29054389
- [Background] Finlayson EV, Birkmeyer JD. Outcomes in vascular surgery: volume versus certification. Surgery. 2001 Nov;130(5):897-8. doi: 10.1067/msy.2001.116926. No abstract available. PMID 11685203
- [Background] Kaplan JA, Finlayson E, Auerbach AD. Impact of Multimodality Pain Regimens on Elective Colorectal Surgery Outcomes. Am Surg. 2017 Apr 1;83(4):414-420. PMID 28424140
- [Background] Oresanya L, Zhao S, Gan S, Fries BE, Goodney PP, Covinsky KE, Conte MS, Finlayson E. Functional outcomes after lower extremity revascularization in nursing home residents: a national cohort study. JAMA Intern Med. 2015 Jun;175(6):951-7. doi: 10.1001/jamainternmed.2015.0486. PMID 25844523
- [Background] Cenzer IS, Tang V, Boscardin WJ, Smith AK, Ritchie C, Wallhagen MI, Espaldon R, Covinsky KE. One-Year Mortality After Hip Fracture: Development and Validation of a Prognostic Index. J Am Geriatr Soc. 2016 Sep;64(9):1863-8. doi: 10.1111/jgs.14237. Epub 2016 Jun 13. PMID 27295578
- [Background] Brembo EA, Kapstad H, Van Dulmen S, Eide H. Role of self-efficacy and social support in short-term recovery after total hip replacement: a prospective cohort study. Health Qual Life Outcomes. 2017 Apr 11;15(1):68. doi: 10.1186/s12955-017-0649-1. PMID 28399883
- [Background] Tang VL, Sudore R, Cenzer IS, Boscardin WJ, Smith A, Ritchie C, Wallhagen M, Finlayson E, Petrillo L, Covinsky K. Rates of Recovery to Pre-Fracture Function in Older Persons with Hip Fracture: an Observational Study. J Gen Intern Med. 2017 Feb;32(2):153-158. doi: 10.1007/s11606-016-3848-2. Epub 2016 Sep 7. PMID 27605004
- [Background] Chereau N, Chandeze MM, Tantardini C, Tresallet C, Lefevre JH, Parc Y, Menegaux F. Antroduodenectomy with Gastroduodenal Anastomosis: Salvage Emergency Surgery for Complicated Peptic Ulcer Disease--Results of a Double Institution Study of 35 Patients. J Gastrointest Surg. 2016 Mar;20(3):539-45. doi: 10.1007/s11605-015-3050-6. Epub 2015 Dec 7. PMID 26643299
- [Background] Ryff CD. In the eye of the beholder: views of psychological well-being among middle-aged and older adults. Psychol Aging. 1989 Jun;4(2):195-201. doi: 10.1037//0882-7974.4.2.195. PMID 2789747
- [Background] Kata A, Sudore R, Finlayson E, Broering JM, Ngo S, Tang VL. Increasing Advance Care Planning Using a Surgical Optimization Program for Older Adults. J Am Geriatr Soc. 2018 Oct;66(10):2017-2021. doi: 10.1111/jgs.15554. Epub 2018 Oct 5. PMID 30289968
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Lawrence VA, Hazuda HP, Cornell JE, Pederson T, Bradshaw PT, Mulrow CD, Page CP. Functional independence after major abdominal surgery in the elderly. J Am Coll Surg. 2004 Nov;199(5):762-72. doi: 10.1016/j.jamcollsurg.2004.05.280. PMID 15501119
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Kraemer HC, Mintz J, Noda A, Tinklenberg J, Yesavage JA. Caution regarding the use of pilot studies to guide power calculations for study proposals. Arch Gen Psychiatry. 2006 May;63(5):484-9. doi: 10.1001/archpsyc.63.5.484. PMID 16651505
- [Derived] Tang V, Pepic L, Higuchi E, Keny C, Macias Lopez E, Onyema EC, Sandhu H, Yank V, Raue PJ. Implementing PST in older adults facing major surgery: a randomised controlled pilot study. BMJ Open. 2025 Nov 12;15(11):e103605. doi: 10.1136/bmjopen-2025-103605. PMID 41224294